CLINICAL TRIAL: NCT01729130
Title: A Pilot Study to Identify the Differences in Adipose Tissue Function After Restoring Normal Glycemic Control Following Pancreas Transplantation
Brief Title: Adipose Tissue Function After Pancreas Transplantation
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 09-043
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; End Stage Renal Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — adipose tissue blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1 Pancreas/kidney transplant: Group 1 of patients with End Stage Renal Disease (ESRD) and Diabetes Mellitis who will receive a pancreas and kidney transplant. An adipose tissue biopsy and blood samples are collected at time of transplant surgery. A repeat adipose tissue needle biopsy and blood samples are collected between 3-12 months post transplant.
  Interventions: Procedure: Adipose tissue biopsy
- Group 2 DM with kidney transplant: Group 2 are patient with DM and ESRD and who will receive only a kidney transplant.
  Interventions: Procedure: Adipose tissue biopsy
- Group 3 No DM and kidney transplant: Group 3 will be patients who do not have DM but do have the diagnosis of ESRD and will receive only a kidney transplant.
  Interventions: Procedure: Adipose tissue biopsy

INTERVENTIONS:
Procedure: Adipose tissue biopsy — Adipose tissue biopsy is done at time of transplant surgery. There is a second needle biopsy done between 3-12 months post transplant surgery.

SUMMARY:
Clinical measures of adipose tissue mass (BMI, waist circumference, waist-to-hip ratio) do not adequately explain the inter-individual and ethnic heterogeneity in diabetes. . There is a need to identify novel/universal markers of risk for diabetes (DM) and cardiovascular disease (CVD). These biomarkers also can become additional outcome measures for an intervention such as pancreatic/kidney transplant. If biological markers show an improvement with an intervention before anthropometric changes occur, intermediate outcomes can be an encouraging finding for practitioners. This study will focus on the central question of "adipose tissue dysfunction" as mediator of metabolic complications of positive energy balance, independent of body fat content and distribution. This study will address the question of effect of hyperglycemia on adipose tissue function independent of body fat mass. This project will take advantage of unique expertise of our investigators to perform detailed metabolic studies in patients with diabetes who undergo pancreatic/kidney transplant. The results of the proposed study will provide support to the novel approach of identifying adipose tissue dysfunction, rather than obesity and fat distribution, as predictor of diabetes and CVD across all ethnic groups, age and gender. We will obtain necessary preliminary data for future grant submissions to support our central hypothesis and develop stronger interactions within and outside The University of Texas Medical Branch (UTMB) with clinical investigators in the area of DM and its complications.

DETAILED DESCRIPTION:
detailed description is his protocol

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of any ethnicity, and age between 18 and 65 years.
2. Patients with diabetes and renal failure who have been scheduled kidney-pancreas or isolated kidney transplantation.
3. Ability to speak read and understand English or Spanish

Exclusion Criteria:

1. Any evidence of acute or severe cardiopulmonary, thyroid, neurological disorders, as assessed by history and physical examination and laboratory testing.
2. Any personal history of substance abuse (reported only).
3. Alcohol intake above 7 grams/day.
4. Pregnancy or lactation.
5. Inability to give consent for this study.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have Diabetes mellitis and End Stage Renal Disease who will be receiving pancreas/kidney or only kidney transplantation.
  Patients that have End Stage Renal Disease and who will be receiving an isolated kidney transplant. This control group will account for effects of immuno-suppression and for potential metabolic changes induced by the kidney transplant on adipose tissue function.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Change in body fat distribution | 1 year post transplantation
  skinfold thickness changes from baseline to within 1 year post transplantation using tape measure, scale and calipers

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cicalese, MD, Principal Investigator — UTMB
Locations (1):
- The University of Texas Medical Branch (UTMB), Galveston, Texas, United States